CLINICAL TRIAL: NCT00991029
Title: Platelet-Oriented Inhibition in New TIA and Minor Ischemic Stroke (POINT) Trial
Acronym: POINT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was halted by the DSMB.
Sponsor: University of California, San Francisco (Other)
Collaborators: Neurological Emergencies Treatment Trials Network (NETT) (Network); Medical University of South Carolina (Other); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1U01S062835-01A1
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Ischemic Attack, Transient
Keywords: Transient Ischemic Attack; TIA; minor stroke
MeSH Terms: conditions — Ischemic Attack, Transient | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- clopidogrel (Active Comparator): Patients assigned to clopidogrel in addition to aspirin
  Interventions: Drug: Clopidogrel
- placebo (Placebo Comparator): Patients assigned to placebo in addition to aspirin
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Clopidogrel — Loading dose of 600mg followed by 75 milligrams, oral, one tablet daily for 89 days
  Other Names: Plavix
  Arms: clopidogrel
Drug: placebo — Loading dose of 8 tablets followed by one tablet daily for 89 days
  Arms: placebo

SUMMARY:
A transient ischemic attack (TIA) is a transient episode of neurological dysfunction caused by focal brain, spinal cord, or retinal ischemia, without acute infarction. An ischemic stroke is a cerebral infarction. In POINT, eligibility is limited to brain TIAs and to minor ischemic strokes (with an NIH Stroke Scale [NIHSS] score less than or equal to 3).

TIAs are common [25], and are often harbingers of disabling strokes. Approximately 250,000-350,000 TIAs are diagnosed each year in the US. Given median survival of more than 8 years [32], there are approximately 2.4 million TIA survivors. In a national survey, one in fifteen of those over 65 years old reported a history of TIA [33], which is equivalent to a prevalence of 2.3 million in older Americans. Based on the prevalence of undiagnosed transient neurological events, the true incidence of TIA may be twice as high as the rates of diagnosis [33]. Based on our review of the National Inpatient Sample for 1997-2003, there were an average of 200,000 hospital admissions for TIA each year, with annual charges climbing quickly in the period to $2.6 billion in 2003.

Composite endpoint of new ischemic vascular events: ischemic stroke, myocardial infarction or ischemic vascular death at 90 days.

DETAILED DESCRIPTION:
Platelet-Oriented Inhibition in New TIA and minor ischemic stroke (POINT) Trial, is a prospective, randomized, double-blind, multicenter trial with the primary null hypothesis that, in patients with TIA or minor ischemic stroke treated with aspirin 50-325 mg/day, there is no difference in the event-free survival at 90 days in those treated with clopidogrel (600 mg loading dose then 75 mg/day) compared to placebo when subjects are randomized within 12 hours of time last known free of new ischemic symptoms.

Its primary objective is to determine whether clopidogrel 75 mg/day by mouth after a loading dose of 600 mg of clopidogrel is effective in preventing major ischemic vascular events (ischemic stroke, myocardial infarction, and ischemic vascular death) at 90 days when initiated within 12 hours of TIA or minor ischemic stroke onset in patients receiving aspirin 50-325 mg/day (with a dose of 150-200 mg daily for 5 days followed by 75-100 mg daily strongly recommended).

Patients over 18 years of age with high-risk TIA (defined as an ABCD2 score greater than or equal to 4) or minor ischemic stroke (with NIHSS less than or equal to 3) who can be treated within 12 hours of time last known free of new ischemic symptoms will be enrolled.

Subjects will be randomized 1:1 (clopidogrel: placebo), controlling for clinical center. A study participant's eligibility will be determined by site personnel prior to accessing the Randomization Module in the WebDCU™, a web-enabled clinical trials management system that was developed by the NETT Statistics and Data Management Center (SDMC) at Medical University of South Carolina (MUSC).Qualified users will access the Randomization Interface and complete a protocol-specific eligibility checklist. If the Randomization Interface finds the patient to be eligible based on the information provided, a randomization number and a confirmatory e-mail are generated.

Each subject is followed for 90 days from randomization; the trial will be completed in 7 years.

A total of 5,840 patients will be recruited. Recruitment will occur over 90 months, with a goal rate of 0.40 subjects/site/month for US sites, and a goal rate of 0.47 subjects/site/month for OUS sites. Current participating sites can be found at: http://www.pointtrial.org/node/18.

ELIGIBILITY:
Inclusion Criteria:

* Neurological deficit (based on history or exam) attributed to focal brain ischemia and EITHER:

  * High risk TIA: Complete resolution of the deficit at the time of randomization AND ABCD2 score of (greater than or equal to) 4 OR
  * Minor ischemic stroke: residual deficit with NIHSS of (less than or equal to) 3 at the time of randomization
* Ability to randomize within 12 hours of time last known free of new ischemic symptoms.
* Head CT or MRI ruling out hemorrhage or other pathology, such as vascular malformation, tumor, or abscess, that could explain symptoms or contraindicate therapy.
* Ability to tolerate aspirin at a does of 50-325 mg/day.

Exclusion Criteria

* Age <18 years
* TIA symptoms limited to isolated numbness, isolated visual changes, or isolated dizziness/vertigo.
* In the judgment of the treating physician, a candidate for thrombolysis, endarterectomy or endovascular intervention, unless the subject declines both endarterectomy and endovascular intervention at the time of evaluation for eligibility.
* Receipt of any intravenous or intra-arterial thrombolysis within 1 week prior to index event.
* Gastrointestinal bleed or major surgery within 3 months prior to index event.
* History of nontraumatic intracranial hemorrhage.
* Clear indication for anticoagulation (e.g., warfarin, heparin) anticipated during the study period (atrial fibrillation, mechanical heart valve, deep venous thrombosis, pulmonary embolism, antiphospholipid antibody syndrome, hypercoagulable state).
* Qualifying ischemic event induced by angiography or surgery.
* Severe non-cardiovascular comorbidity with life expectancy <3 months.
* Contraindication to clopidogrel or aspirin.

  * Known allergy
  * Severe renal (serum creatinine >2 mg/dL or 176.8umol/L) or hepatic insufficiency (prior or concurrent diagnosis, with International Normalized Ratio (INR)>1.5 or any resultant complication, such as variceal bleeding, encephalopathy, or icterus)
  * Hemostatic disorder or systemic bleeding in the past 3 months
  * Current thrombocytopenia (platelet count <100 x10^9/l) or neutropenia (<1 x10^9/l)
  * History of drug-induced hematologic or hepatic abnormalities
* Anticipated requirement for long-term (>7 day) non-study antiplatelet drugs (eg, dipyridamole, clopidogrel, ticlopidine), or Non-steroidal Anti-inflammatory Drugs (NSAIDs) affecting platelet function (such as prior vascular stent or arthritis).
* Inability to swallow medications.
* At risk for pregnancy: premenopausal or post menopausal woman within 12 months of last menses without a negative pregnancy test or not committing to adequate birth control (e.g., oral contraceptive, two methods of barrier birth control, or abstinence).
* Unavailability for follow-up.
* Signed and dated informed consent not obtained from patient.
* Other neurological conditions that would complicate assessment of outcomes during follow-up.
* Ongoing treatment in another study of an investigational therapy that may potentially interact with study drug, or treatment in such a study within the last 7 days.
* Previously enrolled in the POINT study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4881 (Actual)
Dates: Start 2010-05-28 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Claiborne Johnston, MD, PhD, Principal Investigator — University of Texas at Austin; J. Donald Easton, MD, Principal Investigator — University of California, San Francisco; Anthony S. Kim, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (210):
- United States (147):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Banner University Medical Center - Tucson Campus, Tucson, Arizona
  - Mercy San Juan Medical Center, Carmichael, California
  - UCSD Health La Jolla, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Desert Regional Medical Center, Palm Springs, California
  - Huntington Memorial Hospital, Pasadena, California
  - UC Davis Medical Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Scripps Mercy Hospital San Diego, San Diego, California
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - University of Colorado Hospital, Aurora, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Anthony Hospital, Lakewood, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - George Washington University Hospital, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - the Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Evanston Hospital, Evanston, Illinois
  - NorthShore Glenbrook Hospital, Glenview, Illinois
  - Presence Saint Joseph Medical Center, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Southern Illinois University Memorial Medical Center, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - St. Elizabeth Medical Center South, Edgewood, Kentucky
  - St. Elizabeth Hospital, Florence, Kentucky
  - St. Elizabeth Hospital Fort Thomas, Fort Thomas, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Detroit Receiving Hospital, Detroit, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center Hospital, Minneapolis, Minnesota
  - Mayo Clinic Saint Mary's Campus, Rochester, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Mercy Hospital, Springfield, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Benefis Hospitals Inc, Great Falls, Montana
  - Great Falls Clinic Hospital, Great Falls, Great Falls, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - JFK Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - New York Presbyterian / Columbia University Medical Center, New York, New York
  - NYP Weill Cornell Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Strong Memorial Hospital, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Akron City Hospital, Akron, Ohio
  - Mercy Health West Hospital, Cincinnati, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Jewish Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University Hospital, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Pennsylvania State Hershey Medical Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - Vanderbilt University Hospital, Nashville, Tennessee
  - University Medical Center Brackenridge, Austin, Texas
  - Seton Medical Center, Austin, Texas
  - Texas Health Presbyterian Hospital - Dallas, Dallas, Texas
  - Valley Baptist Medical Center - Harlingen, Harlingen, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - UVA Medical Center, Charlottesville, Virginia
  - Bon Secours St. Francis Medical Center, Richmond, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - Henrico Doctors' Hospital - Forest Campus, Richmond, Virginia
  - Henrico Doctors' Hospital - Parham Campus, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - WVU Healthcare Ruby Memorial Hospital, Morgantown, West Virginia
  - Columbia St. Mary's Hospital, Milwaukee, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Australia (9):
  - Gosford Hospital, Gosford, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - The Northern Hospital, Epping, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (9):
  - University of Calgary - Foothills Campus, Calgary, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
  - Charles LeMoyne Hospital, Greenfield Park, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Notre-Dame Hospital, Montreal, Quebec
  - Enfant-Jesus Hospital, Québec
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Turku University Hospital, Turku
- France (6):
  - Fleyriat Hospital, Bourg-en-Bresse
  - Pierre Wetheimer Hospital, Bron
  - Adolphe de Rothschild Ophthalmologic Foundation, Paris
  - Bichat-Claude Bernard Hospital, Paris
  - Pitie-Salpetriere Hospital, Paris
  - Foch Hospital, Suresnes
- Germany (12):
  - University Hospital of Ulm, Ulm, Baden-Wurttemberg
  - Neurological Clinic Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Hospital Neukolln, Berlin
  - Central Bremen Hospital, Bremen
  - University Hospital Essen, Essen
  - University Hospital Frankfurt, Frankfurt
  - University Medical Center Hamburg, Hamburg
  - Hannover Medical School, Hanover
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Schleswig-Holstein Kiel Campus, Kiel
  - University Medical Center Leipzig, Leipzig
  - University Hospital Munster, Münster
- Mexico (5):
  - Mexican Association for Clinical Research, Pachuca, Hidalgo
  - Central Hospital Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí
  - Culiacan General Hospital, Culiacán, Sinaloa
  - Neurosciences Clinical Trials, Culiacán, Sinaloa
  - ABC Medical Center Santa Fe, Mexico City
- Auckland City Hospital, Auckland, New Zealand
- Spain (9):
  - Hospital del Mar, Barcelona
  - Santa Creu and Sant Pau Hospital, Barcelona
  - Vall d'Hebron Hospital, Barcelona
  - Basurto Hospital, Bilbao
  - Burgos University Hospital, Burgos
  - Hospital Donostia, Donostia / San Sebastian
  - Girona University HOspital, Girona
  - La Fe University Hospital, Valencia
  - Miguel Servet Hospital, Zaragoza
- United Kingdom (10):
  - Addenbrooke's Hospital, Cambridge
  - Queen Elizabeth University Hospital, Glasgow
  - Northwick Park Hospital, Harrow
  - The Royal London Hospital, London
  - University College Hospital, London
  - Luton and Dunstable University Hospital, Luton
  - John Radcliffe Hospital, Oxford
  - Royal United Hospital - Bath, Somerset
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent

REFERENCES:
- [Background] Ovbiagele B. Antiplatelet therapy in management of transient ischemic attack: overview and evidence-based rationale. J Emerg Med. 2008 May;34(4):389-96. doi: 10.1016/j.jemermed.2007.08.056. Epub 2008 Jan 18. PMID 18207691
- [Background] Giles MF, Rothwell PM. Risk of stroke early after transient ischaemic attack: a systematic review and meta-analysis. Lancet Neurol. 2007 Dec;6(12):1063-72. doi: 10.1016/S1474-4422(07)70274-0. Epub 2007 Nov 13. PMID 17993293
- [Background] Kernan WN, Schindler JL. Rapid intervention for TIA: a new standard emerges. Lancet Neurol. 2007 Nov;6(11):940-1. doi: 10.1016/S1474-4422(07)70249-1. No abstract available. PMID 17928271
- [Background] Rothwell PM. Transient ischaemic attacks: time to wake up. Heart. 2007 Aug;93(8):893-4. doi: 10.1136/hrt.2007.121111. PMID 17639101
- [Background] Streifler JY. Early stroke risk after a transient ischemic attack: can it be minimized? Stroke. 2008 Jun;39(6):1655-6. doi: 10.1161/STROKEAHA.107.510248. Epub 2008 Mar 27. No abstract available. PMID 18369165
- [Background] Dean N, Shuaib A. Transient ischaemic attacks: unstable, treatable, neglected. Lancet. 2007 Oct 20;370(9596):1398-400. doi: 10.1016/S0140-6736(07)61449-4. No abstract available. PMID 17928045
- [Background] Kennedy J, Hill MD, Ryckborst KJ, Eliasziw M, Demchuk AM, Buchan AM; FASTER Investigators. Fast assessment of stroke and transient ischaemic attack to prevent early recurrence (FASTER): a randomised controlled pilot trial. Lancet Neurol. 2007 Nov;6(11):961-9. doi: 10.1016/S1474-4422(07)70250-8. Epub 2007 Oct 10. PMID 17931979
- [Background] Geisler T, Zurn C, Paterok M, Gohring-Frischholz K, Bigalke B, Stellos K, Seizer P, Kraemer BF, Dippon J, May AE, Herdeg C, Gawaz M. Statins do not adversely affect post-interventional residual platelet aggregation and outcomes in patients undergoing coronary stenting treated by dual antiplatelet therapy. Eur Heart J. 2008 Jul;29(13):1635-43. doi: 10.1093/eurheartj/ehn212. Epub 2008 May 24. PMID 18503057
- [Background] Lotfi A, Schweiger MJ, Giugliano GR, Murphy SA, Cannon CP; TIMI 22 Investigators. High-dose atorvastatin does not negatively influence clinical outcomes among clopidogrel treated acute coronary syndrome patients--a Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 (PROVE IT-TIMI 22) analysis. Am Heart J. 2008 May;155(5):954-8. doi: 10.1016/j.ahj.2007.12.009. Epub 2008 Feb 19. PMID 18440347
- [Background] Mitsios JV, Papathanasiou AI, Rodis FI, Elisaf M, Goudevenos JA, Tselepis AD. Atorvastatin does not affect the antiplatelet potency of clopidogrel when it is administered concomitantly for 5 weeks in patients with acute coronary syndromes. Circulation. 2004 Mar 23;109(11):1335-8. doi: 10.1161/01.CIR.0000124581.18191.15. Epub 2004 Mar 15. PMID 15023882
- [Background] Riondino S, Petrini N, Donato L, Torromeo C, Tanzilli G, Pulcinelli FM, Barilla F. Effects of rosuvastatin on platelet inhibition by clopidogrel in cardiovascular patients. J Thromb Thrombolysis. 2009 Aug;28(2):151-5. doi: 10.1007/s11239-008-0254-6. Epub 2008 Jul 18. PMID 18636229
- [Background] Saw J, Brennan DM, Steinhubl SR, Bhatt DL, Mak KH, Fox K, Topol EJ; CHARISMA Investigators. Lack of evidence of a clopidogrel-statin interaction in the CHARISMA trial. J Am Coll Cardiol. 2007 Jul 24;50(4):291-5. doi: 10.1016/j.jacc.2007.01.097. Epub 2007 Jul 10. PMID 17659194
- [Background] Saw J, Steinhubl SR, Berger PB, Kereiakes DJ, Serebruany VL, Brennan D, Topol EJ; Clopidogrel for the Reduction of Events During Observation Investigators. Lack of adverse clopidogrel-atorvastatin clinical interaction from secondary analysis of a randomized, placebo-controlled clopidogrel trial. Circulation. 2003 Aug 26;108(8):921-4. doi: 10.1161/01.CIR.0000088780.57432.43. Epub 2003 Aug 18. PMID 12925453
- [Background] Trenk D, Hochholzer W, Frundi D, Stratz C, Valina CM, Bestehorn HP, Buttner HJ, Neumann FJ. Impact of cytochrome P450 3A4-metabolized statins on the antiplatelet effect of a 600-mg loading dose clopidogrel and on clinical outcome in patients undergoing elective coronary stent placement. Thromb Haemost. 2008 Jan;99(1):174-81. doi: 10.1160/TH07-08-0503. PMID 18217151
- [Background] Johnston SC, Gress DR, Browner WS, Sidney S. Short-term prognosis after emergency department diagnosis of TIA. JAMA. 2000 Dec 13;284(22):2901-6. doi: 10.1001/jama.284.22.2901. PMID 11147987
- [Background] Coutts SB, Eliasziw M, Hill MD, Scott JN, Subramaniam S, Buchan AM, Demchuk AM; VISION study group. An improved scoring system for identifying patients at high early risk of stroke and functional impairment after an acute transient ischemic attack or minor stroke. Int J Stroke. 2008 Feb;3(1):3-10. doi: 10.1111/j.1747-4949.2008.00182.x. PMID 18705908
- [Background] Coutts SB, Simon JE, Eliasziw M, Sohn CH, Hill MD, Barber PA, Palumbo V, Kennedy J, Roy J, Gagnon A, Scott JN, Buchan AM, Demchuk AM. Triaging transient ischemic attack and minor stroke patients using acute magnetic resonance imaging. Ann Neurol. 2005 Jun;57(6):848-54. doi: 10.1002/ana.20497. PMID 15929051
- [Background] Algra A, van Gijn J, Halkes PH, Kappelle LJ, Koudstaal PJ; ESPRIT Study Group. Interpretation of ESPRIT in the FASTER trial. Lancet Neurol. 2008 Mar;7(3):198-9; author reply 199. doi: 10.1016/S1474-4422(08)70030-9. No abstract available. PMID 18275919
- [Background] Lavallee PC, Meseguer E, Abboud H, Cabrejo L, Olivot JM, Simon O, Mazighi M, Nifle C, Niclot P, Lapergue B, Klein IF, Brochet E, Steg PG, Leseche G, Labreuche J, Touboul PJ, Amarenco P. A transient ischaemic attack clinic with round-the-clock access (SOS-TIA): feasibility and effects. Lancet Neurol. 2007 Nov;6(11):953-60. doi: 10.1016/S1474-4422(07)70248-X. PMID 17928270
- [Background] Luengo-Fernandez R, Gray AM, Rothwell PM. Effect of urgent treatment for transient ischaemic attack and minor stroke on disability and hospital costs (EXPRESS study): a prospective population-based sequential comparison. Lancet Neurol. 2009 Mar;8(3):235-43. doi: 10.1016/S1474-4422(09)70019-5. Epub 2009 Feb 4. PMID 19200786
- [Background] Yusuf S, Diener HC, Sacco RL, Cotton D, Ounpuu S, Lawton WA, Palesch Y, Martin RH, Albers GW, Bath P, Bornstein N, Chan BP, Chen ST, Cunha L, Dahlof B, De Keyser J, Donnan GA, Estol C, Gorelick P, Gu V, Hermansson K, Hilbrich L, Kaste M, Lu C, Machnig T, Pais P, Roberts R, Skvortsova V, Teal P, Toni D, VanderMaelen C, Voigt T, Weber M, Yoon BW; PRoFESS Study Group. Telmisartan to prevent recurrent stroke and cardiovascular events. N Engl J Med. 2008 Sep 18;359(12):1225-37. doi: 10.1056/NEJMoa0804593. Epub 2008 Aug 27. PMID 18753639
- [Background] Sacco RL, Diener HC, Yusuf S, Cotton D, Ounpuu S, Lawton WA, Palesch Y, Martin RH, Albers GW, Bath P, Bornstein N, Chan BP, Chen ST, Cunha L, Dahlof B, De Keyser J, Donnan GA, Estol C, Gorelick P, Gu V, Hermansson K, Hilbrich L, Kaste M, Lu C, Machnig T, Pais P, Roberts R, Skvortsova V, Teal P, Toni D, Vandermaelen C, Voigt T, Weber M, Yoon BW; PRoFESS Study Group. Aspirin and extended-release dipyridamole versus clopidogrel for recurrent stroke. N Engl J Med. 2008 Sep 18;359(12):1238-51. doi: 10.1056/NEJMoa0805002. Epub 2008 Aug 27. PMID 18753638
- [Background] Brown RD Jr, Petty GW, O'Fallon WM, Wiebers DO, Whisnant JP. Incidence of transient ischemic attack in Rochester, Minnesota, 1985-1989. Stroke. 1998 Oct;29(10):2109-13. doi: 10.1161/01.str.29.10.2109. PMID 9756590
- [Background] Kissela B, Broderick J, Woo D, Kothari R, Miller R, Khoury J, Brott T, Pancioli A, Jauch E, Gebel J, Shukla R, Alwell K, Tomsick T. Greater Cincinnati/Northern Kentucky Stroke Study: volume of first-ever ischemic stroke among blacks in a population-based study. Stroke. 2001 Jun;32(6):1285-90. doi: 10.1161/01.str.32.6.1285. PMID 11387488
- [Background] Williams GR, Jiang JG, Matchar DB, Samsa GP. Incidence and occurrence of total (first-ever and recurrent) stroke. Stroke. 1999 Dec;30(12):2523-8. doi: 10.1161/01.str.30.12.2523. PMID 10582972
- [Background] Kleindorfer D, Panagos P, Pancioli A, Khoury J, Kissela B, Woo D, Schneider A, Alwell K, Jauch E, Miller R, Moomaw C, Shukla R, Broderick JP. Incidence and short-term prognosis of transient ischemic attack in a population-based study. Stroke. 2005 Apr;36(4):720-3. doi: 10.1161/01.STR.0000158917.59233.b7. Epub 2005 Feb 24. PMID 15731465
- [Background] Edlow JA, Kim S, Pelletier AJ, Camargo CA Jr. National study on emergency department visits for transient ischemic attack, 1992-2001. Acad Emerg Med. 2006 Jun;13(6):666-72. doi: 10.1197/j.aem.2006.01.014. Epub 2006 Apr 11. PMID 16609106
- [Background] Howard G, Toole JF, Frye-Pierson J, Hinshelwood LC. Factors influencing the survival of 451 transient ischemic attack patients. Stroke. 1987 May-Jun;18(3):552-7. doi: 10.1161/01.str.18.3.552. PMID 3590245
- [Background] Shah KH, Kleckner K, Edlow JA. Short-term prognosis of stroke among patients diagnosed in the emergency department with a transient ischemic attack. Ann Emerg Med. 2008 Mar;51(3):316-23. doi: 10.1016/j.annemergmed.2007.08.016. Epub 2007 Oct 25. PMID 18282526
- [Background] Wu CM, McLaughlin K, Lorenzetti DL, Hill MD, Manns BJ, Ghali WA. Early risk of stroke after transient ischemic attack: a systematic review and meta-analysis. Arch Intern Med. 2007 Dec 10;167(22):2417-22. doi: 10.1001/archinte.167.22.2417. PMID 18071162
- [Background] Gladstone DJ, Kapral MK, Fang J, Laupacis A, Tu JV. Management and outcomes of transient ischemic attacks in Ontario. CMAJ. 2004 Mar 30;170(7):1099-104. doi: 10.1503/cmaj.1031349. PMID 15051693
- [Background] Lisabeth LD, Ireland JK, Risser JM, Brown DL, Smith MA, Garcia NM, Morgenstern LB. Stroke risk after transient ischemic attack in a population-based setting. Stroke. 2004 Aug;35(8):1842-6. doi: 10.1161/01.STR.0000134416.89389.9d. Epub 2004 Jun 10. PMID 15192239
- [Background] Eliasziw M, Kennedy J, Hill MD, Buchan AM, Barnett HJ; North American Symptomatic Carotid Endarterectomy Trial Group. Early risk of stroke after a transient ischemic attack in patients with internal carotid artery disease. CMAJ. 2004 Mar 30;170(7):1105-9. doi: 10.1503/cmaj.1030460. PMID 15051694
- [Background] Hill MD, Yiannakoulias N, Jeerakathil T, Tu JV, Svenson LW, Schopflocher DP. The high risk of stroke immediately after transient ischemic attack: a population-based study. Neurology. 2004 Jun 8;62(11):2015-20. doi: 10.1212/01.wnl.0000129482.70315.2f. PMID 15184607
- [Background] Rothwell PM, Giles MF, Flossmann E, Lovelock CE, Redgrave JN, Warlow CP, Mehta Z. A simple score (ABCD) to identify individuals at high early risk of stroke after transient ischaemic attack. Lancet. 2005 Jul 2-8;366(9479):29-36. doi: 10.1016/S0140-6736(05)66702-5. PMID 15993230
- [Background] Lovett JK, Dennis MS, Sandercock PA, Bamford J, Warlow CP, Rothwell PM. Very early risk of stroke after a first transient ischemic attack. Stroke. 2003 Aug;34(8):e138-40. doi: 10.1161/01.STR.0000080935.01264.91. Epub 2003 Jul 10. PMID 12855835
- [Background] Rao SV, Ohman EM, Granger CB, Armstrong PW, Gibler WB, Christenson RH, Hasselblad V, Stebbins A, McNulty S, Newby LK. Prognostic value of isolated troponin elevation across the spectrum of chest pain syndromes. Am J Cardiol. 2003 Apr 15;91(8):936-40. doi: 10.1016/s0002-9149(03)00107-3. PMID 12686331
- [Background] Whisnant JP, Matsumoto N, Elveback LR. Transient cerebral ischemic attacks in a community. Rochester, Minnesota, 1955 through 1969. Mayo Clin Proc. 1973 Mar;48(3):194-8. No abstract available. PMID 4690325
- [Background] Humphrey PR, Marshall J. Transient ischemic attacks and strokes with recovery prognosis and investigation. Stroke. 1981 Nov-Dec;12(6):765-9. doi: 10.1161/01.str.12.6.765. PMID 7303066
- [Background] Putman SF, Adams HP Jr. Usefulness of heparin in initial management of patients with recent transient ischemic attacks. Arch Neurol. 1985 Oct;42(10):960-2. doi: 10.1001/archneur.1985.04060090042011. PMID 4038103
- [Background] Biller J, Bruno A, Adams HP Jr, Godersky JC, Loftus CM, Mitchell VL, Banwart KJ, Jones MP. A randomized trial of aspirin or heparin in hospitalized patients with recent transient ischemic attacks. A pilot study. Stroke. 1989 Apr;20(4):441-7. doi: 10.1161/01.str.20.4.441. PMID 2648650
- [Background] Dennis M, Bamford J, Sandercock P, Warlow C. Prognosis of transient ischemic attacks in the Oxfordshire Community Stroke Project. Stroke. 1990 Jun;21(6):848-53. doi: 10.1161/01.str.21.6.848. PMID 2349586
- [Background] Coull AJ, Lovett JK, Rothwell PM; Oxford Vascular Study. Population based study of early risk of stroke after transient ischaemic attack or minor stroke: implications for public education and organisation of services. BMJ. 2004 Feb 7;328(7435):326. doi: 10.1136/bmj.37991.635266.44. Epub 2004 Jan 26. PMID 14744823
- [Background] Daffertshofer M, Mielke O, Pullwitt A, Felsenstein M, Hennerici M. Transient ischemic attacks are more than "ministrokes". Stroke. 2004 Nov;35(11):2453-8. doi: 10.1161/01.STR.0000144050.90132.8e. Epub 2004 Oct 14. PMID 15486333
- [Background] Whitehead MA, McManus J, McAlpine C, Langhorne P. Early recurrence of cerebrovascular events after transient ischaemic attack. Stroke. 2005 Jan;36(1):1; author reply 1. doi: 10.1161/01.str.0000149929.92356.f1. No abstract available. PMID 15618448
- [Background] Correia M, Silva MR, Magalhaes R, Guimaraes L, Silva MC. Transient ischemic attacks in rural and urban northern Portugal: incidence and short-term prognosis. Stroke. 2006 Jan;37(1):50-5. doi: 10.1161/01.STR.0000195209.26543.8f. Epub 2005 Dec 1. PMID 16322498
- [Background] Purroy F, Molina CA, Montaner J, Alvarez-Sabin J. Absence of usefulness of ABCD score in the early risk of stroke of transient ischemic attack patients. Stroke. 2007 Mar;38(3):855-6; author reply 857. doi: 10.1161/01.STR.0000257306.00512.d3. Epub 2007 Jan 18. No abstract available. PMID 17234986
- [Background] Wang Y, Johnston SC; CHANCE Investigators. Rationale and design of a randomized, double-blind trial comparing the effects of a 3-month clopidogrel-aspirin regimen versus aspirin alone for the treatment of high-risk patients with acute nondisabling cerebrovascular event. Am Heart J. 2010 Sep;160(3):380-386.e1. doi: 10.1016/j.ahj.2010.05.017. PMID 20826243
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Derived] Balali P, Easton JD, Johnston SC, Cucchiara B. Time to treatment and disability attributed to index stroke in the POINT trial. J Stroke Cerebrovasc Dis. 2024 Nov;33(11):107988. doi: 10.1016/j.jstrokecerebrovasdis.2024.107988. Epub 2024 Sep 1. PMID 39222701
- [Derived] Daghlas I, Johnston SC, Easton JD, Kim AS. Baseline Stroke Risk and Efficacy of Dual-Antiplatelet Therapy: A Post Hoc Analysis of the POINT Trial. Stroke. 2024 Feb;55(2):385-391. doi: 10.1161/STROKEAHA.123.044927. Epub 2024 Jan 4. PMID 38174567
- [Derived] Diener HC, Easton JD, Hart RG, Kasner S, Kamel H, Ntaios G. Review and update of the concept of embolic stroke of undetermined source. Nat Rev Neurol. 2022 Aug;18(8):455-465. doi: 10.1038/s41582-022-00663-4. Epub 2022 May 10. PMID 35538232
- [Derived] Mac Grory B, Piccini JP, Yaghi S, Poli S, De Havenon A, Rostanski SK, Weiss M, Xian Y, Johnston SC, Feng W. Hyperglycemia, Risk of Subsequent Stroke, and Efficacy of Dual Antiplatelet Therapy: A Post Hoc Analysis of the POINT Trial. J Am Heart Assoc. 2022 Feb;11(3):e023223. doi: 10.1161/JAHA.121.023223. Epub 2022 Jan 19. PMID 35043692
- [Derived] Meschia JF, Walton RL, Farrugia LP, Ross OA, Elm JJ, Farrant M, Meurer WJ, Lindblad AS, Barsan W, Ching M, Gentile N, Ross M, Nahab F, Easton JD, Kim AS, Zurita KG, Cucchiara B, Johnston SC. Efficacy of Clopidogrel for Prevention of Stroke Based on CYP2C19 Allele Status in the POINT Trial. Stroke. 2020 Jul;51(7):2058-2065. doi: 10.1161/STROKEAHA.119.028713. Epub 2020 Jun 17. PMID 32568642
- [Derived] Kamel H, Zhang C, Kleindorfer DO, Levitan EB, Howard VJ, Howard G, Soliman EZ, Johnston SC. Association of Black Race With Early Recurrence After Minor Ischemic Stroke or Transient Ischemic Attack: Secondary Analysis of the POINT Randomized Clinical Trial. JAMA Neurol. 2020 May 1;77(5):601-605. doi: 10.1001/jamaneurol.2020.0010. PMID 32091536
- [Derived] Cucchiara B, Elm J, Easton JD, Coutts SB, Willey JZ, Biros MH, Ross MA, Johnston SC. Disability After Minor Stroke and Transient Ischemic Attack in the POINT Trial. Stroke. 2020 Mar;51(3):792-799. doi: 10.1161/STROKEAHA.119.027465. Epub 2020 Feb 12. PMID 32078486
- [Derived] Farrant M, Easton JD, Adelman EE, Cucchiara BL, Barsan WG, Tillman HJ, Elm JJ, Kim AS, Lindblad AS, Palesch YY, Zhao W, Pauls K, Walsh KB, Marti-Fabregas J, Bernstein RA, Johnston SC. Assessment of the End Point Adjudication Process on the Results of the Platelet-Oriented Inhibition in New TIA and Minor Ischemic Stroke (POINT) Trial: A Secondary Analysis. JAMA Netw Open. 2019 Sep 4;2(9):e1910769. doi: 10.1001/jamanetworkopen.2019.10769. PMID 31490536
- [Derived] Johnston SC, Elm JJ, Easton JD, Farrant M, Barsan WG, Kim AS, Lindblad AS, Palesch YY, Zurita KG, Albers GW, Cucchiara BL, Kleindorfer DO, Lutsep HL, Pearson C, Sethi P, Vora N; POINT and Neurological Emergencies Treatment Trials Network Investigators. Time Course for Benefit and Risk of Clopidogrel and Aspirin After Acute Transient Ischemic Attack and Minor Ischemic Stroke. Circulation. 2019 Aug 20;140(8):658-664. doi: 10.1161/CIRCULATIONAHA.119.040713. Epub 2019 Jun 26. PMID 31238700
- [Derived] Tillman H, Johnston SC, Farrant M, Barsan W, Elm JJ, Kim AS, Lindblad AS, Palesch YY, Easton JD. Risk for Major Hemorrhages in Patients Receiving Clopidogrel and Aspirin Compared With Aspirin Alone After Transient Ischemic Attack or Minor Ischemic Stroke: A Secondary Analysis of the POINT Randomized Clinical Trial. JAMA Neurol. 2019 Jul 1;76(7):774-782. doi: 10.1001/jamaneurol.2019.0932. PMID 31034032
- [Derived] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Derived] Zhao W, Pauls K. Architecture design of a generic centralized adjudication module integrated in a web-based clinical trial management system. Clin Trials. 2016 Apr;13(2):223-33. doi: 10.1177/1740774515611889. Epub 2015 Oct 13. PMID 26464429
- [Derived] Johnston SC, Easton JD, Farrant M, Barsan W, Battenhouse H, Conwit R, Dillon C, Elm J, Lindblad A, Morgenstern L, Poisson SN, Palesch Y. Platelet-oriented inhibition in new TIA and minor ischemic stroke (POINT) trial: rationale and design. Int J Stroke. 2013 Aug;8(6):479-83. doi: 10.1111/ijs.12129. PMID 23879752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clopidogrel | Placebo
Started | 2432 | 2449
Completed | 2276 | 2281
Not Completed | 156 | 168

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel | Placebo | Total
Number analyzed (Participants) | 2432 | 2449 | 4881
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at time of randomization
  years | 65.0 [55.0 to 74.0] | 65.0 [56.0 to 74.0] | 65.0 [55.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1097 | 1098 | 2195
  Male | 1335 | 1351 | 2686
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Race or ethnic group was determined by the investigator. Hispanic ethnic group was assessed only in patients in the United States.
  Participants
    Hispanic or Latino | 144 | 146 | 290
    Not Hispanic or Latino | 2176 | 2182 | 4358
    Unknown or Not Reported | 112 | 121 | 233
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 16 | 23
  Asian | 77 | 67 | 144
  Native Hawaiian or Other Pacific Islander | 10 | 5 | 15
  Black or African American | 473 | 493 | 966
  White | 1774 | 1781 | 3555
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 87 | 82 | 169
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 3 | 4 | 7
  Canada | 121 | 119 | 240
  United States | 2014 | 2029 | 4043
  Finland | 25 | 25 | 50
  Mexico | 5 | 4 | 9
  United Kingdom | 33 | 38 | 71
  Australia | 53 | 51 | 104
  France | 51 | 47 | 98
  Germany | 8 | 10 | 18
  Spain | 119 | 122 | 241
Qualifying Event [Count of Participants; unit: Participants] — TIA or Ischemic Stroke
  Participants
    TIA | 1056 | 1052 | 2108
    Ischemic Stroke | 1376 | 1397 | 2773
Qualifying Neurologic Score [Median (Inter-Quartile Range); unit: units on a scale] — The ABCD2 score is a seven-point score for identifying patients who have suffered a transient ischemic attack (TIA) at the highest risk of stroke (scores ranges from 0 to 7, with higher scores indicating a greater risk of stroke).
  The National Institutes of Health Stroke Scale (NIHSS) score is used quantify the impairment caused by a stroke (scores range from 0 to 42, with higher scores indicating greater stroke severity).
  Patients were eligible if they had an acute ischemic stroke with a score of 3 or less on the NIHSS or had a TIA with a score of 4 or more on the ABCD2 scale. Population: ABCD2 scores were available for 2104 of the 2108 patients with TIA (1055 patients in the clopidogrel group and 1049 in the placebo group). NIHSS scores were available for 2750 of the 2773 patients with ischemic stroke (1365 patients in the clopidogrel group and 1385 in the aspirin group).
  units on a scale
    ABCD2: number analyzed (Participants) | 1055 | 1049 | 2104
    ABCD2 | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 5.0] | 5.0 [4.0 to 6.0]
    National Institutes of Health Stroke Scale: number analyzed (Participants) | 1365 | 1385 | 2750
    National Institutes of Health Stroke Scale | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]

OUTCOME MEASURES:

1. Primary Outcome: Composite of Ischemic Stroke, Myocardial Infarction, or Death From Ischemic Vascular Causes
Description: Primary efficacy outcome: Number of Participants with Ischemic Stroke, Myocardial Infarction, or Death From Ischemic Vascular Causes
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 121 | 160
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.02, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.59 to 0.95]

2. Primary Outcome: Major Hemorrhage
Description: Primary safety outcome: Number of Participants with major hemorrhage
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 23 | 10
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.02, Log Rank; Hazard Ratio (HR) = 2.32, 95% CI 2-sided [1.10 to 4.87]

3. Secondary Outcome: Ischemic Stroke
Description: Secondary efficacy outcome:Number of participants with Ischemic stroke
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 112 | 155
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.01, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.56 to 0.92]

4. Secondary Outcome: Myocardial Infarction
Description: Secondary efficacy outcome: Number of participants with Myocardial infarction
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 10 | 7
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.46, Log Rank; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.55 to 3.78]

5. Secondary Outcome: Death From Ischemic Vascular Causes
Description: Secondary efficacy outcome: Number of participants with Death from ischemic vascular causes
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 6 | 4
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.52, Log Rank; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.43 to 5.35]

6. Secondary Outcome: Ischemic or Hemorrhagic Stroke
Description: Secondary efficacy outcome: Number of participants with Ischemic or hemorrhagic stroke
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 116 | 156
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.01, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.94]

7. Secondary Outcome: Composite of Ischemic Stroke, Myocardial Infarction, Death From Ischemic Vascular Causes, or Major Hemorrhage
Description: Secondary efficacy outcome: Number of participants with ischemic stroke, myocardial infarction, death from ischemic vascular causes, or major hemorrhage
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 141 | 167
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.13, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.05]

8. Other Pre Specified Outcome: Hemorrhagic Stroke
Description: Other safety outcome: Number of participants with Hemorrhagic stroke
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 5 | 3
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.47, Log Rank; Hazard Ratio (HR) = 1.68, 95% CI 2-sided [0.4 to 7.03]

9. Other Pre Specified Outcome: Symptomatic Intracerebral Hemorrhage
Description: Other safety outcome: Number of participants with Symptomatic intracerebral hemorrhage
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 2 | 2
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.99, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.14 to 7.14]

10. Other Pre Specified Outcome: Other Symptomatic Intracranial Hemorrhage
Description: Other safety outcome: Number of participants with other symptomatic intracranial hemorrhage
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 2 | 0
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.16, Log Rank

11. Other Pre Specified Outcome: Major Hemorrhage Other Than Intracranial Hemorrhage
Description: Other safety outcome: Number of Participants with Major hemorrhage other than intracranial hemorrhage
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 17 | 7
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.04, Log Rank; Hazard Ratio (HR) = 2.45, 95% CI 2-sided [1.01 to 5.9]

12. Other Pre Specified Outcome: Minor Hemorrhage
Description: Other safety outcome:Number of Participants with Minor hemorrhage
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 40 | 13
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 3.12, 95% CI 2-sided [1.67 to 5.83]

13. Other Pre Specified Outcome: Death From Any Cause
Description: Other safety outcome: Number of Participants with Death from any cause
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 2432 | 2449
Participants | 18 | 12
Statistical Analysis 1: Comparison: Clopidogrel vs Placebo; Test type: Superiority; p = 0.27, Log Rank; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.73 to 3.13]

ADVERSE EVENTS:
Time Frame: 90 days from randomization
Description: Only serious adverse events or protocol-defined clinical outcomes were collected (not all non-serious adverse events). The clinical outcomes also have been reported under the outcomes section.
  Some, but not all, non-serious adverse events were collected and they are included in the 'Other (not including serious) Adverse Events' table below.
Arm/Group | Clopidogrel | Placebo
All-Cause Mortality (participants affected / at risk) | 18/2432 | 12/2449
Serious Adverse Events (participants affected / at risk) | 382/2432 | 382/2449
Other Adverse Events (participants affected / at risk) | 89/2432 | 84/2449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=2432) | Placebo (N=2449)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Arterial repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspiration bronchial (Investigations) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 24 (24) | 15 (15)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
Atrial septal defect (Congenital, familial and genetic disorders) | 2 (2) | 2 (2)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiomyopathy acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 10 (10) | 17 (17)
Carotid artery stent insertion (Surgical and medical procedures) | 0 (0) | 2 (2)
Carotid body tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 7 (7) | 7 (8)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 18 (18) | 22 (24)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 13 (13) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 1 (1) | 1 (1)
Complicated migraine (Nervous system disorders) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1) | 3 (3)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 9 (10) | 10 (10)
Coronary artery disease (Cardiac disorders) | 4 (4) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 5 (5)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Drug rehabilitation (Surgical and medical procedures) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 5 (5) | 0 (0)
Endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 (11) | 1 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 3 (3) | 3 (3)
Haemorrhagic transformation stroke (Nervous system disorders) | 4 (4) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3)
Hypertensive crisis (Vascular disorders) | 1 (1) | 6 (6)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Implant site haemorrhage (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-cerebral aneurysm operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 3 (3) | 4 (4)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 82 (83) | 113 (118)
Lacunar infarction (Nervous system disorders) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Meningitis leptospiral (Infections and infestations) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 4 (4) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 4 (5)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 5 (5)
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1) | 2 (2)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 3 (3)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Somatisation disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 6 (6) | 4 (4)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 49 (54) | 55 (62)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=2432) | Placebo (N=2449)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral amyloid angiopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 4 (4)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 7 (7) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 4 (4) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 13 (14) | 19 (19)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 40 (43) | 42 (46)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT00991029/SAP_000.pdf
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT00991029/Prot_001.pdf